CLINICAL TRIAL: NCT03735251
Title: Epidemic Profile of Left Ventricular Diastoic Dysfunction in the Community Elderly and Establishing Prediction Model: the Northern Shanghai Study
Acronym: ELITISM
Status: Completed | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Shanghai 10th People's Hospital, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: ELITISM
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2014-07

CONDITIONS: Left Ventricular Diastoic Dysfunction Cohort Study
Keywords: Left Ventricular Diastoic Dysfunction Cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Venous blood samples are obtained after an overnight fast. Total cholesterol, high-density lipoprotein cholesterol and triglycerides are measured by standard methods, and the Friedewald formula is used to calculate the lowdensity lipoprotein (LDL) cholesterol (LDL-c). Other biological parameters like plasma/urine albumin and creatinine are measured by standard methods at local laboratories. The urine albumin-to-creatinine ratio (UACR) is also calculated. The serum and urine samples will be stored at -80°C. Prior to storage, the date, number of vials and recorder's name will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left Ventricular Diastoic Dysfunction Classification: normal diastole pattern：E/A>1，DT 160~220 ms，S/D >1，AR 0.22-0.32m/sec，E/e'< 8 diastolic dysfunction pattern Impaired relaxation pattern：E/A< 1，DT > 220 ms，S/D > 1，AR 0.21-0.28 m/sec，E/e'<10 Pseudo-normalization pattern：E/A> 1，DT 150~210 ms，S/D < 1，AR ≥0.35m/sec，E/e'≥ 10 Restrictive pattern：E/A ≥ 2，DT < 150 ms，S/D <1，AR ≥0.25m/sec，E/e'≥10
  Interventions: Other: Diuretic，Betaloc，antiplatelet drugs

INTERVENTIONS:
Other: Diuretic，Betaloc，antiplatelet drugs — According to international guidelines,we treated patinets who suffered from different disease

SUMMARY:
This study is one of the largest ongoing prospective population studies to evaluate target organ damages (TODs) and Left Ventricular Diastoic Dysfunction in the community-dwelling elderly Chinese, which is authorised and funded by the Shanghai municipal government.This study was approved by the Shanghai Tenth People's Hospital Institutional Review Board and was conducted under financial support from the Shanghai municipal government (grant ID: 2013ZYJB0902 and 15GWZK1002). The preliminary sample size is expected to be 3000-4000 participants.

DETAILED DESCRIPTION:
The Northern Shanghai Study is an ongoing prospective community-based study. After enrolment, clinical examination,anthropometric measurement and a questionnaire will be administered to each participant at baseline and patients will be followed up every six months. Our tests and examinations include: blood/urine sample and biochemical measurements, office blood pressure recording, carotid ultrasonograph, echocardiograph, pulse wave velocity, pulse wave analysis, 4-limb blood pressure recording, body mass index, etc. Baseline measurement will also include the assessments on target organ damages(TODs) and the conventional CV risk factors. In the follow-up, the incidence of CV events and mortality will be recorded. The Northern Shanghai Risk Score will be calculated, with considerations on CV risk factors and TODs.

ELIGIBILITY:
Inclusion Criteria:

1. age 55 years or more
2. informed consent should be signed voluntarily
3. local residents from communities in northern Shanghai and available for long-term follow-up

Exclusion Criteria:

1. was diagnosed with serious heart disease (NYHA≥IV) or end-stage renal disease (CKD ≥4 stage)
2. suffered from cancer or his/her life expectancy is <5 years
3. had stroke within 3 months
4. is not willing to participate in the clinical study
5. has to quit the trial due to other diseases
6. violates the protocol or loses contact with the laboratory staff.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Northern Shanghai region has the largest population of elderly adults in Shanghai, with a total population of 1.57 million and an elderly proportion of over 19%. We use a computer-generated list of communities, and 10 communities were randomly selected for the first-phase enrolment. Other communities in the list will be randomly selected for the later enrolment. According to the inclusion and exclusion criteria, we invite all the eligible older people (over 55 years) to participate in this study. The recruitment strategies include: (1) posting study recruitment files in the neighbourhood committees and community hospitals; (2) according to the health file, community hospitals recruit the potential participants Open Accessby telephone; (3) hand out recruitment flyers directly to the potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 1920 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2014-08-10 (Actual)

PRIMARY OUTCOMES:
left ventricular diastolic dysfunction | From July 2014 to August 2019
  All the ultrasonography measurements are performed with a MyLab 30 CV machine (ESAOTE SpA, Genoa, Italy), according to the American Society of Echocardiography (ASE) recommendations.The echocardiography is performed in the left decubitus position. Left ventricular (LV) internal diameter at end-diastole (LVIDd) and septal (SWTd) and posterior wall thickness at end-diastole (PWTd) are measured directly.
  left ventricular diastolic dysfunction including: Impaired relaxation pattern：E/A< 1，DT > 220 ms，S/D > 1，AR 0.21-0.28 m/sec，E/e'<10 Pseudo-normalization pattern：E/A> 1，DT 150~210 ms，S/D < 1，AR ≥0.35m/sec，E/e'≥ 10 Restrictive pattern：E/A ≥ 2，DT < 150 ms，S/D <1，AR ≥0.25m/sec，E/e'≥10